CLINICAL TRIAL: NCT00726102
Title: Development and Health of Rural Chinese Children Fed Meat as a Daily Complementary Food From 6-18 Mos of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Xi-Chou Women and Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-0768; Thrasher
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Nutritional Deficiencies
Keywords: Zinc nutrition; Growth; Development; China; Infants; Toddlers
MeSH Terms: conditions — Malnutrition | interventions — Meat; Edible Grain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meat (Active Comparator): Provide locally available meat daily to infants from 6 to 18 mos of age
  Interventions: Other: Meat
- Control (Active Comparator): Daily provision of cereal to infants from 6-18 mos
  Interventions: Other: Cereal
- Fortified rice cereal (Active Comparator): Provide equi-caloric serving of fortified rice cereal on daily basis from 6-18 months of age
  Interventions: Other: fortified rice cereal

INTERVENTIONS:
Other: Meat — 2 0z of locally available meat per day
  Arms: Meat
Other: Cereal — Daily provision of cereal to infants from 6-18 mos
  Arms: Control
Other: fortified rice cereal — Daily provision of fortified cereal to infants 6-18 months of age
  Arms: Fortified rice cereal

SUMMARY:
Inadequate feeding of infants and toddlers impairs physical and cognitive development and is a major contributor to early childhood infectious disease illnesses and preventable mortality. Optimal feeding has two broad components: Exclusive breast feeding (EBF) for the first-6 months followed by continued breast feeding accompanied by complementary foods (CF) that is adequate in quantity and quality. While EBF is theoretically straightforward, CF is more complex. This is because CF is typically limited mainly or entirely to plant-based foods in developing countries worldwide. Dependence on adequate, affordable locally-produced foods for complete CF requires an inexpensive, regular source of meat especially to provide 'problem' micronutrients, notably, but not only, zinc and bioavailable iron. While the use of micronutrient-fortified CF and of supplements, including SprinklesTM, is spreading, their efficacy largely remains uncertain as does their availability, particularly on a sustainable, affordable basis Achievement of the widespread regular use of meat as a CF requires: (1) adequate local production of affordable small scavenging/foraging animals in poor rural and, where feasible, periurban communities worldwide; (2) effective communication for behavioral change/education so that young children, starting at age 6 months (when meat is readily accepted by infants), receive priority in the use of this meat. Solid scientific evidence of the value of international/national programs to achieve this goal is essential to provide the basis and incentive for major international and national programs to promote the feeding of meat as an early and regular CF. The acquisition of such evidence is the goal of this study

The intervention to be evaluated is meat fed daily as a complementary food from age 6-18 months. Thirty infants-toddlers in each of 60 rural communities (total of 1,800 subjects) will participate. In a cluster design, twenty communities (test) will be randomized to receive meat,twenty communities (control) will receive a plant recipe providing the same amount of calories, twenty communities (fortified cereal) will receive a commercially available fortified cereal providing the same amount of calories. This project will be located in rural China in a county where high quality collaboration is already established, and where we have recently demonstrated inadequate bioavailable zinc intake and zinc deficiency in toddlers. We have also found a high (30%) incidence of stunting, now widely used as an indirect indicator of populations with zinc deficiency. Other advantages of this location include the willingness of doctors located in each rural community to provide the test or control meal 7 days per week in their homes and the absence of any access to supplements / fortified products which could complicate interpretation of data. The young children in the test communities will receive certified safe lean pork 7 days per wk. Starting with a very small quantity at 6 months, the quantity of lean pork will be increased as infants are ready to take more up to a plateau of 2 oz/d. No subsequent increases are planned because neither zinc nor iron requirements increase from 6-11 months to 12-18 months. Lean pork will be used because pigs are ubiquitous in China and can be maintained cheaply by scavenging/foraging on waste materials adjacent to human habitation. Test and control clusters will also receive nutrition education to achieve maximal diversification of locally available affordable foods. Longitudinal outcome measures include indices of physical growth, especially length; infectious disease incidence and prevalence; cognitive development; zinc and iron intake and biomarkers for these and other micronutrients. Zinc absorption will be measured. Data will flow daily from communities to the district hospital in Xi-Chou, weekly to the data manager in Shanghai and 3-monthly to the Data Monitoring Safety Board (DSMB) and to the University of Colorado research group.

DETAILED DESCRIPTION:
Objectives The goal of this project is to determine the efficacy of a daily intake of locally available, low cost meat as a complementary food for young children aged 6-18 months who are otherwise dependent on continued breast feeding and locally available non-fortified plant foods only. Efficacy will be determined by public health outcomes, including infectious disease morbidity and both physical and cognitive development, with linear growth as the primary outcome measure. Other outcome measures required for interpretation of these results are food and nutrient intake; biomarkers of key micronutrient status; zinc absorption and measures of host factor that might compromise the effects of optimizing nutrition.

Rationale Inadequate complementary feeding (CF) is a major contributor to preventable morbidity and mortality in young children in the developing world. Except in emergency situations, inadequate macronutrient intake is largely attributable to lack of adequate maternal knowledge, while optimal micronutrient intake depends on food diversity. Though food fortification programs can diminish or possibly eradicate the need for food diversity, reliable sources of affordable fortified foods/supplements are frequently unavailable and their efficacy not always certain. Locally grown, nutritionally complete affordable sources of CF are and will remain a key strategy especially for the millions of rural poor. Adequate food diversity depends on meat to provide adequate zinc and also a favorable source of bioavailable iron, in addition to assuring sufficient intake of other key micronutrients, e.g. vitamin B12. Meat's theoretical benefits in CF have not, however, been tested adequately. Clear demonstration of public health benefits is essential to support policies to promote local production of adequate, affordable small foraging animals with priority use for older infants/toddlers. The long-term goal is to achieve nutritionally complete complementary feeding from affordable local sources for millions of poor rural/semi-rural young children worldwide.

Methods The project is an unmasked randomized controlled trial with cluster design in which 60 rural village communities, each with 30 infants, within the County of Xi-Chou, Wen-Shan, Yunnan Province, SW China will be randomly selected and randomly assigned to intervention or control clusters. The intervention will be meat fed daily from age 6-18 months. Control participants will receive an equi-caloric rice-based supplement or a commercially available fortified rice cereal. The intervention team will include 80 community doctors, supervised and supported by senior staff at Xi-Chou Women's and Children's Hospital. This senior staff will be also be responsible for purchasing and quality of intervention foods. The intervention meat will be certified safe pork, because pigs are ubiquitous in rural China and can be maintained cheaply by foraging/scavenging. Lean pork, which will be increased as accepted up to a plateau of 2 oz/d, will be provided as a meat-rice recipe daily in the community doctors' homes; any food remaining will be fed at home later in the day. Control children will receive a daily plant-based recipe or fortified rice cereal also in their community doctors' homes. Starting at the time of recruitment at age 3 months, monthly nutrition education messages will be given to mothers. Initially focusing on exclusive breast feeding; after 6 months of age, education for both test and control clusters will focus on optimizing diversity of locally available, affordable complementary foods and on responsive feeding (messages designed to increase energy intake are not required in this population). Specially trained local and Shanghai health research teams will obtain longitudinal outcome measures between 6-18 months. Outcomes include: anthropometry at 6, 9, 12, 15 and 18 months; daily records of infectious disease morbidity (kept by community doctors); Bayley Scales of Infant Development III at 6, 12, 18 months plus the WHO motor questionnaire; 24-hr dietary recall data at 6, 7, 9, 12, 15 18 months; biomarkers and, on a subsample, measurements of zinc absorption and gut function at 6, 9 and 18 months. Data will be transferred daily to the local research base at Xi-Chou Women and Children's Hospital, checked for accuracy and entered into the data management system. These data will be transferred weekly to the data manager in Shanghai Jiao Tong University, School of Medicine, Xin-Hua Hospital. Data will be collated and shared with the Colorado research group at 3-monthly intervals. SAS software will be used for a range of outcome-specific statistical measures.

Significance Positive outcomes for meat group versus controls will provide scientific justification for promotion of production of affordable small animal meats globally in rural/semi-rural and even peri-urban communities and of communication for behavioral change/education to provide meat as a regular complementary feed from age 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 3 months of age

Exclusion Criteria:

* birth wt <2000 g
* any chronic disease or condition that affects growth
* not breastfed

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1488 (Actual)
Dates: Start 2008-11; Primary Completion 2012-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Linear Growth | 6-18 mos of age

SECONDARY OUTCOMES:
Morbidity | 6-18 mos of age
Cognitive development | 0-18 mo of age
Zn absorption | 9 and 18 mos of age

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hambidge, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Tang M, Sheng XY, Krebs NF, Hambidge KM. Meat as complementary food for older breastfed infants and toddlers: a randomized, controlled trial in rural China. Food Nutr Bull. 2014 Dec;35(4 Suppl):S188-92. doi: 10.1177/15648265140354S304. PMID 25639137
- [Derived] Sheng X, Wang J, Li F, Ouyang F, Ma J. Effects of dietary intervention on vitamin B12 status and cognitive level of 18-month-old toddlers in high-poverty areas: a cluster-randomized controlled trial. BMC Pediatr. 2019 Sep 13;19(1):334. doi: 10.1186/s12887-019-1716-z. PMID 31519167